CLINICAL TRIAL: NCT02542683
Title: Physical Activity and Cognitive Development in Children
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Lena S. Sun, E.M. Papper Professor of Pediatric Anesthesiology, Columbia University
Other Study IDs: AAAP7626
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Diseases; Children
Keywords: congenital heart diseases; cognition; adaptive behavior; physical activity; neurodevelopment
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Because the blood sampling will only be performed when the study subject will be having his or her routine blood tests either as a part of preoperative testing, or as follow up for his or her clinical condition, there will be no additional discomfort or problems associated with the blood draw.
  The amount of blood we will be asking for the study is approximately 5 ml, of about one teaspoonful. We will test for the following: cytokine panel (Tumor necrosis factor(TNF-alpha), Interleukins (IL-1ß, IL-6, IL-8), CRP and other relevant biomarkers as indicated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- physical activity program: enrollment for 12 months in a structured physical activity program
  Interventions: Other: structured physical activity program
- delayed physical activity program: No intervention for 12 months, then enrollment in structured physical activity program

INTERVENTIONS:
Other: structured physical activity program — a structured modest physical activity program
  Groups: physical activity program

SUMMARY:
1. Compare physical activity and cognitive functions between children having cardiac surgery with an age-matched group of children undergoing non-cardiac surgery, as well as otherwise healthy siblings or best buddies (or age and gender-matched children if no siblings or best buddies available) before surgery and after surgery or six months following initial assessment.
2. Determine the effects of a structured physical activity program for 6 months following surgery on cognitive functions and adaptive behavior in children following congenital cardiac surgery.
3. Determine the effects of a structured physical activity program for 12 months following surgery on cognitive functions and adaptive behavior in children following congenital cardiac surgery.
4. We will perform exploratory analysis to determine whether any effects of a 12-months structured physical activity program on cognitive functions and adaptive behavior persist beyond 12 months after cessation of the program.

DETAILED DESCRIPTION:
Mortality associated with congenital heart defects (CHD) has decreased significantly world-wide over the past decades. As more CHD patients are surviving beyond infancy and childhood, these patients are found to be at significant risk for developmental disabilities and developmental delay. In CHD patients, their neurodevelopmental impairments, as suggested by recent data from the Boston Circulatory Arrest Trial, appear to become more serious with increasing age. As they mature into adolescents and adults, more areas of neurocognitive abnormalities become evident. These abnormalities significantly influence their ability to function independently in their daily living and impact their quality of life. Physical activity has been shown to improve cognitive function in adults and improve attentional inhibition and cognitive flexibility in school-age children between 7 to 9 years of age. An exercise program has also been shown to improve self-reported cognitive functioning and parent-reported social functioning in older children and adolescents (age 10-25 years) with Tetralogy of Fallot or single ventricle physiology. Of note, neuroimaging studies have further documented that physical activity induces an increase in hippocampal volume which corresponds to the observed improvement in memory tasks. Since neurocognitive functions in CHD patients become worse as they get older, any early intervention that can mitigate the neurocognitive impairment in these patients will modify their negative neurodevelopmental trajectory and thus could have a major impact on the mental and cognitive well-being of CHD patients. The purpose of our study is to test the hypothesis that a regular, structured physical activity program as recommended by the American Heart Association will improve cognitive function and adaptive behavior in children with CHD after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Diseases (CHD) Cohort: All children with congenital cyanotic cardiac diseases scheduled for congenital cardiac surgery who are older than 30 months of age.
* Non-CHD, Surgical Cohort: All children 30 months or older who are undergoing non-cardiac surgery at Columbia University Medical Center (CUMC), including pediatric general surgery, urological surgery, ear, nose and throat (ENT) surgery, plastic surgery and eye surgery. These children will be recruited before surgery.
* Non-surgical cohort:

  1. Sibling of children of CHD patients within 12 months in age, and 30 months of age or older.
  2. Relatives of CHD patients of the same gender within 12 months in age and 30 months of age or older.
  3. Best buddies of CHD children within 12 months in age and 30 months of age or older.
  4. Children who are matched by age ±6 months who are 30 months of age or older, gender, level parental education and language spoken at home

Exclusion Criteria:

1. Children with known chromosomal syndromes, or known syndromes including but not limited to DiGeorge, Trisomy 21, WIlliams, Noonan and Turner.
2. Children with known physical disabilities.
3. Children with known history of central nervous system (CNS) injury including stroke, birth asphyxia, seizure disorder, intraventricular hemorrhage.
4. Children with abnormal neurological exam by a pediatric physician or nurse practitioner, and confirmed by a pediatric neurologist.
5. Children with tricuspid regurgitation on echocardiography or on cardiac angiography that is moderate or greater.
6. Children with moderate or greater decrease in ventricular function on echocardiography or on cardiac angiography.
7. Children with baseline room air oxygen saturation below 80%.
8. Children who are treated for dysrhythmias or are pacemaker-dependent.
9. Children with history of prematurity. (Non-surgical cohort)
10. Children with history of more than one episode of hospitalization. (Non-surgical cohort)

Ages: 30 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Physicians or nurse practitioner who are providers of care for CHD patients from the pediatric cardiology and/or cardiothoracic surgical services will make initial contact with parents of potential study subjects regarding enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Intelligence Quotient (IQ) score | Up to 24 months from the time of assessment at baseline
  Global neurocognitive function assessment with IQ score using the Wechsler Preschool and Primary Scale of Intelligence (WPPSI 4): at baseline and up to 24 months later.
Score on the NIH Toolbox Early Childhood Battery | Up to 24 months from the time of assessment at baseline
  Domain-specific neurocognitive function: Memory, learning, attention, executive function, language and motor function using the NIH Toolbox Early Childhood. Scores from each domain in the battery will be used . Domain-specific scores obtained at baseline, then every 6 months up to 24 months later.
Score on Adaptive Behavior Assessment System, 3rd edition (ABAS-III) | Up to 24 months from the time of assessment at baseline
  Adaptive behavior: Parental reports of behavior using ABAS-III, collected at baseline and then every 6 months up to 24 months later.

SECONDARY OUTCOMES:
Weight | Up to 24 months from baseline
  Record weight and plot on growth curve at baseline, then every 6 months for 18 months.
Height | Up to 24 months from baseline
  Record height and plot on growth curve at baseline, then every 6 months for 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lena S. Sun, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No